CLINICAL TRIAL: NCT01853852
Title: A Phase I, Randomized, Single-Blind, Four-Period Cross-Over, Placebo-Controlled, Dose-Escalation Study to Evaluate the Safety and Pharmacokinetics of Single Oral Doses of GR181413A/AT1001 in Healthy Japanese Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Amicus Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single
Other Study IDs: 115806
Record Dates: First submitted 2011-11-10; First posted 2013-05-15 (Estimated); Last update posted 2013-12-18 (Estimated); Status verified 2013-12

CONDITIONS: Fabry Disease
MeSH Terms: conditions — Fabry Disease | interventions — migalastat; larazotide acetate; Drinking Water

STUDY DESIGN:
Who Masked: Participant

ARMS (4):
- 50 mg (Experimental): GR181413A/AT1001
  Interventions: Drug: GR181413A/AT1001 solution; Other: Potable water; Drug: Placebo capsule
- 150 mg (Experimental): GR181413A/AT1001
  Interventions: Drug: GR181413A/AT1001 capsule
- 450 mg (Experimental): GR181413A/AT1001
  Interventions: Drug: GR181413A/AT1001 capsule
- Placebo (Placebo Comparator): placebo
  Interventions: Drug: GR181413A/AT1001 solution; Drug: GR181413A/AT1001 capsule; Other: Potable water; Drug: Placebo capsule

INTERVENTIONS:
Drug: GR181413A/AT1001 solution — Powder for reconstitution
  Arms: 50 mg; Placebo
Drug: GR181413A/AT1001 capsule — Size 2, hard gelatin capsule, white opaque / blue opaque
  Arms: 150 mg; 450 mg; Placebo
Other: Potable water — Matched, Size 2, hard gelatin capsule, white opaque/blue opaque
  Arms: 50 mg; Placebo
Drug: Placebo capsule — Solution matched
  Arms: 50 mg; Placebo

SUMMARY:
GR181413A/AT1001 (migalastat hydrochloride) is a low molecular weight iminosugar, an analog of the terminal galactose group that is cleaved from the substrate GL-3. This compound was researched and developed as a drug for treatment of Fabry disease. This study, MGM115806, will be the first administration of GR181413A/AT1001 to Japanese subjects to investigate the safety, tolerability and pharmacokinetics of single oral doses in healthy Japanese adult subjects. Approximately 12 subjects will receive three treatments of 50, 150 and 450 mg GR181413A/AT1001 under fasted conditions plus placebo in a dose ascending crossover design. Serial pharmacokinetic samples will be collected and safety assessments will be performed following each dose. The pharmacokinetics and dose proportionality of GR181413A/AT1001 after single oral doses of GR181413A/AT1001 at the dose levels of 50, 150 and 450 mg under fasted conditions will be assessed.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy as determined by a responsible and experienced physician, based on a medical evaluation including medical history, physical examination, laboratory tests and cardiac monitoring. A subject with a clinical abnormality or laboratory parameters outside the reference range for the population being studied may be included only if the Investigator and the GSK Medical Monitor agree that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures.
2. Male or female between 20 and 55 years of age inclusive, at the time of signing the informed consent.
3. A female subject is eligible to participate if she is of: Non-childbearing potential defined as pre-menopausal female.
4. Male subjects with female partners of child-bearing potential must agree to use one of the contraception methods. This criterion must be followed from the time of the first dose of study medication until 5 terminal half-lives post-last dose.
5. Body weight >=50 kg and BMI within the range 18.5 - 29.0 kg/m2 (inclusive).
6. Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.
7. AST, ALT, alkaline phosphatase and bilirubin > 1.5xULN (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%).
8. Single QTcB or QTcF < 450 msec; or QTc < 480 msec in subjects with Bundle Branch Block.
9. Japanese defined being born in Japan, having four ethnic Japanese grandparents, holding a Japanese passport or identity papers and being able to speak Japanese. Japanese subjects should be also have lived outside Japan for less than 10 years.

Exclusion Criteria:

1. A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of screening.
2. A positive pre-study drug/alcohol screen.
3. A positive test for HIV antibody.
4. History of regular alcohol consumption within 6 months of the study
5. The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longest).
6. Exposure to more than four new chemical entities within 12 months prior to the first dosing day.
7. Use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements (including St Johns Wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study medication, unless in the opinion of the Investigator and GSK Medical Monitor the medication will not interfere with the study procedures or compromise subject safety.
8. History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or GSK Medical Monitor, contraindicates their participation.
9. Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 56 day period.
10. History or regular use of tobacco- or nicotine-containing products within 6 months prior to screening.
11. Pregnant females as determined by positive serum or urine hCG test at screening or prior to dosing.
12. Lactating females.
13. Unwillingness or inability to follow the procedures outlined in the protocol.
14. Subject is mentally or legally incapacitated.

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2011-09; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Profile of plasma pharmacokinetics | 0, 0.5, 1, 1.5, 2, 3, 3.5, 4, 5, 6, 8, 10, 12h post dose
  AUC, Cmax, tmax, Tlast , t1/2, CL/F, Vz/F
Number of Participants with adverse events | up to 24 hr
Change from baseline in clinical laboratory tests (hematology, chemistry and urinalysis) | 0, 24h post dose
Change from baseline in vital signs (blood pressure and heart rate) | 0 ,1 , 2, 3, 4, 5, 6, 24h post dose
Change from baseline in 12-lead ECG | 0, i, 2, 3, 6, 24h post dose
Profile of urine pharmacokinetics | 0-4, 4-10, 10-12, 12-24h post dose
  Ae, CLr, %Fx

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Clinical Research, Study Director — Amicus Therapeutics
Locations (1):
- GSK Investigational Site, Randwick, New South Wales, Australia

REFERENCES:
- [Derived] Ino H, Takahashi N, Terao T, Mudd PN Jr, Hirama T. Pharmacokinetics, safety, and tolerability following single-dose migalastat hydrochloride (GR181413A/AT1001) in healthy male Japanese subjects. J Drug Assess. 2013 Jul 24;2(1):87-93. doi: 10.3109/21556660.2013.827117. eCollection 2013. PMID 27536442